CLINICAL TRIAL: NCT03243305
Title: AMPOWER A Single-arm, Phase III, Open Label, Multi-center, Study in Women Aged 18-35 Years of the Contraceptive Efficacy and Safety of Phexxi™ (Previously Referred to as AMPHORA®) Contraceptive Vaginal Gel
Brief Title: AMP002 Phase III Contraceptive Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Evofem Inc. (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AMP002
Record Dates: First submitted 2017-06-29; First posted 2017-08-09 (Actual); Results first posted 2020-07-22 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Contraception

STUDY DESIGN:
Intervention Model Description: Single Arm, unblinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): This is a single-arm, open-label, Phase III study of AMPHORA , a non-hormonal contraceptive, at approximately 100 sites in the United States (US) over seven cycles of use in women aged 18 to 35 years who are at risk of pregnancy.
  Interventions: Drug: AMPHORA

INTERVENTIONS:
Drug: AMPHORA — non-hormonal contraceptive vaginal gel

SUMMARY:
This is a single-arm, open-label, Phase III study in approximately 100 sites in the United States (US) over seven cycles of use in women aged 18 to 35 years who are at risk of pregnancy.

DETAILED DESCRIPTION:
Through assessments including pelvic examination, laboratory procedures, and medical and gynecological history, subjects will be screened for eligibility in order to enroll approximately 1349 subjects into the study. After a screening period of up to 60 days, enrolled women will receive study drug. Each woman will participate in the study until after she has completed treatment during seven study cycles. Women who have individual cycles that do not meet the criteria for an evaluable cycle will not have those cycles replaced by subsequent cycles in order to provide a total of seven evaluable cycles.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

To enroll in the clinical study, potential subjects must:

1. Be healthy women, who are sexually active, at risk of pregnancy, and desiring contraception.
2. Be within the age range of 18 to 35 years old (inclusive) at enrollment.
3. In the opinion of the Investigator, be at low risk for both human immunodeficiency virus (HIV) and sexually transmitted infections (STIs) based on review of high-risk behaviors and exposures according to the Centers for Disease Control STI Guideline.
4. At the time of enrollment, have a single male sex partner for ≥3 months.
5. Have a negative urine pregnancy test at enrollment.
6. Have normal, cyclic menses with a usual length of 21 to 35 days over the last two cycles or at least two consecutive spontaneous menses (21 to 35 days in length) since delivery, abortion, or after discontinuing hormonal contraception or hormonal therapy prior to the date of consent. In addition:

   1. If the subject recently discontinued breastfeeding, she must have demonstrated return to regular cycling and have had at least three consecutive, spontaneous menses post-lactation prior to the date of consent.
   2. If the subject received prior administration of injectable contraceptives (e.g., depot-medroxyprogesterone acetate [DMPA], Depo Provera), there must be at least 10 months since the last injection and the subject must have had at least two consecutive, spontaneous menses prior to the date of consent.
   3. If a contraceptive implant was recently removed, the subject must have had at least two consecutive, spontaneous menses prior to the date of consent.
   4. If an intrauterine device (IUD) was recently removed, the subject must have had at least one spontaneous menses following removal and prior to the date of consent.
7. Be willing to engage in at least three acts of heterosexual vaginal intercourse per cycle.
8. Be willing to use the study drug as the only method of contraception over the course of the study (with the exception of emergency contraception [EC] in the event a subject engages in vaginal intercourse but believes that the study drug was not used properly or she is at risk for pregnancy for any other reason).
9. Be capable of using the study drug properly and agree to comply with all study directions and requirements, including retaining the wrappers and returning them to the clinical site at the next study visit.
10. Be willing to keep a daily electronic diary (eDiary) to record coital information, study drug use information, use of concomitant medications including other vaginal products and other contraceptives, menses, and sign and symptom data for the subject or as reported to her by her partner.
11. Agree not to participate in any other clinical studies during the course of the study.
12. Be capable and willing to give written informed consent to participate in the study.

Exclusion Criteria:

Exclusion Criteria:

To enroll in the clinical study, potential subjects must not:

1. Have had three or more urinary tract infections (UTIs) in the past year from the date of consent.
2. Have a UTI by urine culture, chlamydia, gonorrhea, or symptomatic yeast vaginitis or symptomatic bacterial vaginosis (BV) diagnosed by wet mount, or trichomoniasis, unless treated and proof of cure is documented within the screening period.
3. Have used vaginal or systemic antibiotics or antifungals within 14 days prior to enrollment, with the exception of vaginal or systemic antibiotics or antifungals completed for the treatment of a UTI, BV, or yeast vaginitis diagnosed at screening within seven days of the Enrollment Visit.
4. Have a history of any recurrent vaginal infections/disorders (either greater than or equal to four times in the past year or greater than or equal to three times in the previous six months from the date of consent).
5. Be pregnant, have a suspected pregnancy, or desire to become pregnant during the course of the study.
6. Have a history of diagnosed infertility or of conditions that may lead to infertility, without subsequent non-assisted reproductive technology intrauterine pregnancy.
7. Have any maternal contraindications to pregnancy (medical condition) or chronic use of medications for which significant evidence of fetal risk exists.
8. Have known or screen test positive for HIV infection.
9. Have three or more outbreaks of genital herpes simplex virus (HSV) within the last year from the date of consent or be receiving suppressive therapy.
10. Have visible genital condylomata (warts).
11. Be lactating or breastfeeding.
12. Have any clinically significant abnormal finding on physical examination including pelvic examination or baseline laboratory assessments which in the opinion of the Investigator, precludes study participation.
13. Have clinically significant signs of vaginal or cervical irritation on pelvic examination.
14. Be planning to have any (e.g., diagnostic or therapeutic) vaginal or cervical procedures during the period of the study.
15. Have an abnormal Papanicolaou test (Pap test) based on the following criteria:

    a. Pap test in the past 12 months from the date of screening with atypical squamous cells of undetermined significance (ASC-US) unless at least one of the following criteria is met: i. Less than 21 years of age. ii. A repeat Pap test at least six months later was normal. iii. Reflex human papillomavirus (HPV) testing was performed and was negative for high-risk HPV.

    iv. A colposcopy (with or without biopsy) found no evidence of dysplasia requiring treatment or treatment was performed and follow up at least six months after the treatment showed no evidence of disease.

    b. Pap test in the past 12 months from the date of screening with low grade squamous intraepithelial lesion (LSIL) unless at least one of the following criteria is met: i. Less than 21 years of age. ii. A colposcopy (with or without biopsy) found no evidence of dysplasia requiring treatment or treatment was performed and follow up at least six months after the treatment showed no evidence of disease.

    c. Pap test in the past 12 months from the date of screening with atypical squamous cells in which high grade squamous intraepithelial lesion cannot be excluded (ASC-H), atypical glandular cells, high grade squamous intraepithelial lesion (HSIL), or ≥30 years old who are cytology negative and HPV 16- or HPV 18-positive unless colposcopy and/or treatment was performed and follow up at least six months after the colposcopy and/or treatment showed no evidence of disease.

    d. Pap test in the past 12 months with malignant cells.
16. Consume (on average) more than three drinks of an alcoholic beverage per day.
17. In the opinion of the Investigator, have a history of substance abuse in the last 12 months.
18. Have taken an investigational drug or used an investigational device within the past 30 days from the date of consent.
19. In the opinion of the Investigator, have issues or concerns that may compromise the safety of the subject, impact the subject's compliance with the protocol requirements, or confound the reliability of the data acquired.
20. Be an Evofem, PAREXEL, or clinical site employee regardless of direct involvement in research activities, or their close relative.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 1384 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2018-11-29 (Actual); Study Completion 2018-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Culwell, Study Director — Evofem Inc.
Locations (87):
- United States (87):
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - East Valley Family Physicians 137, Chandler, Arizona
  - Mesa Obstetricians & Gynecologists 184, Mesa, Arizona
  - Family Practice Specialists Ltd 170, Phoenix, Arizona
  - Precision Trials AZ, LLC 176, Phoenix, Arizona
  - Radiant Research, Inc. 111, Scottsdale, Arizona
  - Visions Clinical Research Tucson 138, Tucson, Arizona
  - Eclipse Clinical Research 185, Tucson, Arizona
  - Arkansas Primary Care Clinic 205, Little Rock, Arkansas
  - Anaheim Clinical Trials, LLC 135, Anaheim, California
  - Essential Access Health 159, Berkeley, California
  - Hope Clinical Research, LLC 163, Canoga Park, California
  - Grossmont Center for Clinical Research 119, La Mesa, California
  - Northern California Research 179, Sacramento, California
  - Medical Center for Clinical Research 101, San Diego, California
  - Optimal Research, LLC 149, San Diego, California
  - Women's Health Care 122, San Diego, California
  - Harbor - UCLA LABIOMED 143, Torrance, California
  - Empire Clinical Research 175, Upland, California
  - Lynn Institute of the Rockies 172, Colorado Springs, Colorado
  - Downtown Women's Healthcare 109, Denver, Colorado
  - Coastal Connecticut Research, LLC 141, New London, Connecticut
  - Flordia Clinical Research Group, LLC 130, Clearwater, Florida
  - Clinical Physiology Associates 160, Fort Myers, Florida
  - AGA Clinical Trials 108, Hialeah, Florida
  - Health Care Family Rehab and Research Center 193, Hialeah, Florida
  - The Community Research of South Florida 167, Hialeah, Florida
  - Vital Pharma Research, Inc. 123, Hialeah, Florida
  - UF Health Woman's Specialist - Emerson 194, Jacksonville, Florida
  - Health Awareness, Inc. 129, Jupiter, Florida
  - Altus Research 142, Lake Worth, Florida
  - Optimal Research, LLC 107, Melbourne, Florida
  - South Florida Research Center, Inc. 165, Miami, Florida
  - Advanced Pharma CR, LLC 156, Miami, Florida
  - AppleMed Research Group, LLC 154, Miami, Florida
  - New Horizon Research 155, Miami, Florida
  - Vista Health Research 166, Miami, Florida
  - Heuermd Research, Inc. 140, Orlando, Florida
  - Health Care Family Rehab and Research 190, Pembroke Pines, Florida
  - Physician Care Clinical Research 158, Sarasota, Florida
  - Visions Clinical Research 168, Wellington, Florida
  - Agile Clinical Research Trials 161, Atlanta, Georgia
  - Atlanta North Gynecology, PC 120, Roswell, Georgia
  - Elite Clinical Trials 105, Blackfoot, Idaho
  - Women's Health Practice 132, Champaign, Illinois
  - American Health Network, Inc. - Avon 144, Avon, Indiana
  - Women's Health Advantage 162, Fort Wayne, Indiana
  - American Health Network, Inc. - Franklin 146, Franklin, Indiana
  - American Health Network, Inc. - Muncie 145, Muncie, Indiana
  - Clinical Trials Management, LLC 131, Covington, Louisiana
  - Frederick OB/GYN 189, Frederick, Maryland
  - ActivMed Practices & Research, Inc. 133, Methuen, Massachusetts
  - Saginaw Valley Medical Research Group, LLC 124, Saginaw, Michigan
  - Planned Parenthood of the St. Louis Regions 169, St Louis, Missouri
  - Office of Edmond Pack, MD 192, Las Vegas, Nevada
  - Clinical Research Center of Nevada 136, Las Vegas, Nevada
  - R. Garn Mabey, Jr., MD, Chartered 116, Las Vegas, Nevada
  - Bosque Women's Care 117, Albuquerque, New Mexico
  - Upstate Clinical Research Associates 114, Williamsville, New York
  - PMG Research of Cary 134, Cary, North Carolina
  - Unified Women's Clinical Research 125, Morehead City, North Carolina
  - Eastern Carolina Women's Center 103, New Bern, North Carolina
  - Lyndhurst Clinical Research 110, Raleigh, North Carolina
  - Southeastern Research Center 139, Winston-Salem, North Carolina
  - Radient Research, Inc. 152, Cincinnati, Ohio
  - Elite Research Network - Rapid Medical Research, Inc. 171, Cleveland, Ohio
  - Aventiv 128, Columbus, Ohio
  - Complete Healthcare for Women 151, Columbus, Ohio
  - Clinical Research of Philadelphia 186, Philadelphia, Pennsylvania
  - Medical Research South 126, Charleston, South Carolina
  - The University of Tennessee Medical Center 188, Knoxville, Tennessee
  - Premier Family Physicians 102, Austin, Texas
  - Pioneer Research Solutions, Inc. 164, Beaumont, Texas
  - Family Medicine Associates of Texas 106, Carrollton, Texas
  - Practice Research Organization 115, Dallas, Texas
  - Brownstone Clinical Trials 191, Fort Worth, Texas
  - Centex Studies, Inc. 182, Houston, Texas
  - Southeast Texas Family Planning & Cancer Screening 121, Houston, Texas
  - Texas Center for Drug Development. Inc. 150, Houston, Texas
  - North Texas Family Medicine 104, Plano, Texas
  - Neera Bhatia, MD OB/GYN 180, San Antonio, Texas
  - Progressive Clinical Research 187, San Antonio, Texas
  - Physician's Research Options, LLC 178, Draper, Utah
  - Wasatch Clinical Research 183, Salt Lake City, Utah
  - PI-Coor Clinical Research, LLC 153, Centreville, Virginia
  - Clinical Research Associates of Tidewater 148, Norfolk, Virginia
  - Seattle Women's: Health, Research, Gynecology 113, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Interventional: This is a single-arm, open-label, Phase III study of AMPHORA, a non-hormonal contraceptive, at 112 sites in the United States (US) over seven cycles of use in women aged 18 to 35 years who are at risk of pregnancy.
  AMPHORA: non-hormonal contraceptive vaginal gel
Period: Overall Study
Arm/Group | Interventional
Started | 1384
Completed | 449
Not Completed | 935
Not completed — Lost to Follow-up | 250
Not completed — Withdrawal by Subject | 170
Not completed — Pregnancy | 104
Not completed — Non-Compliance with Study Drug | 38
Not completed — Adverse Event | 23
Not completed — No sexually active | 26
Not completed — Physician Decision | 22
Not completed — Protocol Violation | 22
Not completed — Study method no longer primary method | 12
Not completed — Study Terminated by Sponsor | 1
Not completed — Early terminations | 267

BASELINE CHARACTERISTICS:
Arm/Group | Interventional
Number analyzed (Participants) | 1384
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.7 (4.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1384
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 571
  Not Hispanic or Latino | 805
  Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6
  Asian | 35
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 348
  White | 955
  More than one race | 0
  Unknown or Not Reported | 38
Body Mass Index (BMI) at Screening [Mean (Standard Deviation); unit: kg/m^2] | 28.770 (8.1079)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Pregnancy Outcomes to Measure Contraceptive Efficacy
Description: To evaluate the contraceptive efficacy of Amphora over 7-cycle of use
Time Frame: 10 months
Population: MITT population that included only those subjects whose diaries indicated that they used the study drug correctly for every act of intercourse for at least 1 menstrual cycle. Cycles in which the study drug was used incorrectly for 1 or more coital acts were removed, and the remaining cycles were aligned in order to provide contiguous cycles.
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional
Number analyzed (Participants) | 1182
Participants | 100
Statistical Analysis 1: Comparison: Interventional; The primary hypothesis to be tested is whether subjects using Amphora vaginal gel have a 7-cycle cumulative pregnancy percentage less than or equal to 21%; Test type: Other; Kaplan-Meier; Seven-cycle Pregnancy Percentage = 13.65, 95% CI 2-sided [9.91 to 17.39]

2. Secondary Outcome: Number of Subjects With Adverse Events (AE)
Description: Incidence of AE to evaluate safety
Time Frame: 10 months
Population: All subjects enrolled into the study and who administered the study drug at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional
Number analyzed (Participants) | 1330
Participants
  Subjects with greater than or equal to 1 AE | 601
  Subjects with greater than or equal to 1 SAE | 17
  AE leading to early discontinuation | 25
  Relationship of AEs: unlikely to be Related | 186
  Relationship of AEs: possibly related | 166
  Relationship of AEs: probably related | 139
  Relationship of AEs: definitely related | 108
  Relationship of AEs: not assessable | 2
  Intensity of AEs: mild | 318
  Intensity of AEs: moderate | 249
  Intensity of AEs: severe | 31
  Intensity of AEs: life-threatening | 3
  Death | 0

ADVERSE EVENTS:
Time Frame: 10 months
Description: An AE was defined as any unfavorable and unintended sign (including abnormal laboratory finding), symptom, or disease temporally associated with the use of the study drug, whether or not it is considered related.
Arm/Group | Interventional
All-Cause Mortality (participants affected / at risk) | 0/1330
Serious Adverse Events (participants affected / at risk) | 17/1330
Other Adverse Events (participants affected / at risk) | 601/1330
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Interventional (N=1330)
Peritoneal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Cystitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Uterine rupture (Injury, poisoning and procedural complications) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Status epilepticus (Nervous system disorders) | 1
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 1
Bipolar I disorder (Psychiatric disorders) | 1
Depression suicidal (Psychiatric disorders) | 1
Vaginal disorder (Reproductive system and breast disorders) | 1
Trisomy 21 (Pregnancy, puerperium and perinatal conditions) | 1 — Pregnancy-related SAEs that were reported after study completion
Preeclampsia (Pregnancy, puerperium and perinatal conditions) | 1 — Pregnancy-related SAEs that were reported after study completion
Premature rupture of membrane (Pregnancy, puerperium and perinatal conditions) | 1 — Pregnancy-related SAEs that were reported after study completion
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Interventional (N=1330)
Bacterial vaginosis (Infections and infestations) | 37
Nasopharyngitis (Infections and infestations) | 35
Urinary tract infection (Infections and infestations) | 76
Vulvovaginal mycotic infection (Infections and infestations) | 38
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 266
Vulvovaginal pain (Reproductive system and breast disorders) | 51
Vulvovaginal pruritus (Reproductive system and breast disorders) | 149

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-11-01): https://cdn.clinicaltrials.gov/large-docs/05/NCT03243305/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-24): https://cdn.clinicaltrials.gov/large-docs/05/NCT03243305/SAP_001.pdf